CLINICAL TRIAL: NCT00050440
Title: A Phase 2 Study of ET-743 as Second-Line Therapy in Subjects With Persistent or Recurrent Endometrial Carcinoma
Brief Title: Phase 2 Study of ET-743 (Trabectedin) in Patients With Persistent or Recurrent Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004429; ET743-USA-1 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); NCT01328314 (obsolete NCT alias)
Record Dates: First submitted 2002-12-09; First posted 2002-12-10 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Endometrial Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female Urogenital Neoplasms
Keywords: Endometrial; Cancer; Carcinoma; Trabectedin; Ecteinascidin 743; ET743; Antineoplastic Agents; Alkylating Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Neoplasms; Carcinoma | interventions — Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin (Experimental): Trabectedin 1.3 mg/m2 administered intravenously every 21 days. Dexamethasone 4 mg administered orally (by mouth) the day before the trabectedin dose, 30 minutes before the trabectedin dose, and for 2 days following the trabectedin dose.
  Interventions: Drug: Trabectedin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Trabectedin — Trabectedin 1.3 mg/m2 administered intravenously every 21 days.
Drug: Dexamethasone — Dexamethasone 4 mg administered orally (by mouth) the day before the trabectedin dose, 30 minutes before the trabectedin dose, and for 2 days following the trabectedin dose

SUMMARY:
The purpose of this is to test the safety and effectiveness of an investigational chemotherapy agent in patients with persistent or recurrent endometrial cancer.

DETAILED DESCRIPTION:
Patients will be enrolled in the study after all study-specific entry criteria are met and informed consent is obtained. Patients will be required to attend regular clinic visits to receive study medication and have their status monitored. They will also be required to have radiologic tumor assessments performed at multiple times throughout the study. A detailed explanation can be provided by the Investigator conducting this study. Trabectedin 1.3 mg/m2 will be given every 21 days to patients intravenously (i.v). over a 3-hour period via a central venous catheter (referred to as a "central line") which is a tube (ie, catheter) placed into a large vein that is used to administer medications. Dexamethasone 4 mg will be given orally (p.o.) the day before trabectedin and dexamethasone 20 mg will be given i.v. 30 minutes before trabectedin. Dexamethasone 4 mg p.o. will be given for 2 days following trabectedin administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or metastatic endometrial carcinoma
* Progressive disease after 1 cytotoxic chemotherapy regimen given for advanced/metastatic disease
* At least one measureable tumor lesion
* Adequate bone marrow, hepatic and renal function
* Performance status ECOG 0 or 1

Exclusion Criteria:

* Prior exposure to trabectedin
* Known hypersensitivity to dexamethasone or to any of the components of trabectedin
* Less than 4 weeks since last radiation therapy or since last dose of hormonal therapy, biological therapy, therapy with any investigational agent, or chemotherapy
* History of another neoplastic disease unless in remission for more than 5 years
* Known metastases (spread) of cancer to the central nervous system or other serious illness as specified in the protocol
* Current pregnancy, lactation, or childbearing potential without adequate method of contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-07; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with objective response | Up to approximately 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 3 years
The number of patients with adverse events | Up to approximately 3 years
Time to progression (TTP) | Up to approximately 3 years
Progression free survival (PFS), | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (14):
- United States (8):
  - Los Angeles, California
  - Miami, Florida
  - Lexington, Kentucky
  - Baltimore, Maryland
  - New York, New York
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Dallas, Texas
- Toronto, Ontario, Canada
- Maastricht, Netherlands
- Russia (4):
  - Moscow
  - Obninsk
  - Saint Petersburg
  - Saint

REFERENCES:
- See also: McMeekin DS, Lisyanskaya A, Crispens M, et al. Single-agent trabectedin as second-line therapy of persistent or recurrent endometrial cancer: results of a multi-center phase II study. Gynecol Oncol. 2009;114(2):288-92. — http://dx.doi.org/10.1016/j.ygyno.2009.04.034